CLINICAL TRIAL: NCT04464109
Title: Comparative Motility of Retro-scleral and Intrascleral Orbital Implants After Evisceration
Brief Title: Comparative Motility of Alloplastic Orbital Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mostafa Mohammed Mohammed Diab, Principal investigator, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R116/2020
Record Dates: First submitted 2020-07-05; First posted 2020-07-09 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Anophthalmos; Acquired; Evisceration; Traumatic, Eye
Keywords: Evisceration; Orbital implant; Implant position; Implant motility
MeSH Terms: conditions — Anophthalmos

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retro-scleral placement of the implant (Active Comparator): Surgical steps;
  1. Two anterior scleral relaxing incisions
  2. A 360° scleral incision around the optic nerve to disinsert it
  3. Two posterior scleral relaxing incisions
  4. The implant is inserted posterior to posterior scleral edges
  5. The posterior sclera is closed then the anterior sclera is overlapped and closed.
  6. The implant is completely seated in the intraconal space
  Interventions: Procedure: Evisceration with orbital implantation
- Intrascleral placement of the implant (Active Comparator): Anterior and posterior sclerotomies with the implant partly in the scleral shell and partly in the intraconal space.
  1. Anterior relaxing sclerotomies not reaching the optic nerve
  2. A 360° scleral incision around the optic nerve.
  3. The anterior sclera flaps are overlapped and closed
  4. Part of the implant remains in the scleral shell, while the remaining part is sitting in the intraconal space.
  Interventions: Procedure: Evisceration with orbital implantation

INTERVENTIONS:
Procedure: Evisceration with orbital implantation — Evisceration will be performed. Alloplastic orbital implant will be inserted either posterior to the sclera or partly within the scleral canal.

SUMMARY:
This study will evaluate the effect of posterior placement of orbital implants on their motility compared to intrascleral placement after evisceration .

DETAILED DESCRIPTION:
Evisceration allows removal of the intraocular contents while preserving the sclera and normal extraocular muscle attachments. It is more advantageous than enucleation in patients in whom intraocular tumor is rules out.

Maximizing orbital volume and restoration of movement are important aspects of a successful surgical outcome.

Standard evisceration techniques do not allow placement of an implant larger than 13-16 mm which don't adequately replace the volume leading to postevisceration socket syndrome. Therefore, various techniques have been described to expand the scleral cavity and allow placement of a large implant including anterior sclerotomies, posterior sclerotomies, and disinsertion of optic nerve.

Implant exposure is a terrible complication of evisceration with reported rates as high as 67%. Exposure of the implant can lead to infection, which usually mandates removal of the implant. Trying to minimize this risk, physicians intentionally place the implants posterior to the normal position of the globe. Some authors described placement of the implant posterior to posterior sclera which totally eliminated the risk of exposure.

However, this deep seating of the implant may have deleterious effects on its motility. It can decrease implant-prosthesis interaction. In addition, retro-scleral placement of the implant moves it posterior to the pulleys that serve as the functional origins of rectus muscles. This relationship would be expected to alter the pulling directions of the rectus muscles after evisceration hindering effective implant motility.

In this trial the investigators will try to study the effect of posterior placement of the implants on its motility after evisceration.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are candidates for evisceration

Exclusion Criteria:

* Inability to provide independent, informed consent
* Significant preoperative motility abnormalities

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Implant motility | 6 months
  The conjunctiva is marked at the center point of the implant while the patient looking in primary gaze. The excursion of the mark will be measured will a standard millimeter ruler in extreme gaze positions
Prosthesis motility | 6 months
  It will be measured with the kestenbaum's limbus test. Photographs will be taken while patients wearing Kestenbaum spectacles in vertical and horizontal directions of gaze.

SECONDARY OUTCOMES:
Volume augmentation | 6 months
  Exophthalmometry will be performed for all patients after fitting a prosthesis. Enophthalmos is to be graded from 1 to 4 (grade 1 = no postoperative improvement; grade 2 = improvement <2 mm but remained enophthalmos; grade 3 = improvement ≥2 mm but remained enophthalmos; and grade 4 = no enophthalmos) compared with unaffected side.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Mohammed M Diab, PhD, Principal Investigator — Fayoum University Hospitals
Locations (1):
- Mostafa Mohammed Mohammed Diab, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available upon reasonable request from the corresponding author, after deidentification. The data are not publicly available due to their containing information that could compromise the privacy of research participants. Study protocol will be also available. Data will be available for researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available beginning 6 months after starting the trial and ending 12 months following article publication
Access Criteria: from corresponding author